CLINICAL TRIAL: NCT04225091
Title: Efficacy Evaluation of Triple up® Collagen Drink on Skin Condition
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: TCI Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 19-098-B
Record Dates: First submitted 2020-01-06; First posted 2020-01-13 (Actual); Last update posted 2020-11-30 (Actual); Status verified 2020-11

CONDITIONS: Skin Condition
MeSH Terms: conditions — Skin Diseases

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo drink (Placebo Comparator)
  Interventions: Dietary Supplement: Blank
- Triple up® Collagen Drink (Experimental)
  Interventions: Dietary Supplement: Testing product

INTERVENTIONS:
Dietary Supplement: Testing product — consume 1 bottle (50 mL) per day for 28 days
  Other Names: Triple up® Collagen Drink
  Arms: Triple up® Collagen Drink
Dietary Supplement: Blank — consume 1 bottle (50 mL) per day for 28 days
  Other Names: Placebo drink
  Arms: Placebo drink

SUMMARY:
To assess Triple up® Collagen Drink on skin condition improvement

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults aged above 20 years old

Exclusion Criteria:

* Subject who is not willing to participate in this study.
* Patients with diseases of the skin, heart, liver, kidney, endocrine and other organs and patients with mental illness (according to medical history).
* Subjects who have known cosmetic, drug or food allergies, difficulty in digestive tract absorption or disorder.
* Female who is pregnant or nursing or planning to become pregnant during the course of the study.
* Received facial laser therapy, chemical peeling or UV overexposure in the past 4 weeks.
* Vegetarian
* Subjects who have large spots (area >3 square centimeter) or abnormal acne.

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2020-01-30 (Actual); Primary Completion 2020-04-21 (Actual); Study Completion 2020-05-07 (Actual)

PRIMARY OUTCOMES:
The change of skin moisture | Change from Baseline skin moisture at 4 weeks
  Corneometer® CM825 was utilized to measure skin moisture. Units: arbitrary Corneometer® units 0-120
The change of skin elasticity | Change from Baseline skin elasticity at 4 weeks
  Cutometer® dual MPA 580 was utilized to measure skin elasticity (parameter R2). Units: μm penetration depth into the probe opening, expressed as curves
The change of skin wrinkles | Change from Baseline skin wrinkles at 4 weeks
  VISIA Complexion Analysis System was utilized to measure wrinkles. Units: arbitrary units
The change of skin collagen density | Change from Baseline skin collagen density at 4 weeks
  DermaLab® USB - 20 MHz High Freq. Ultrasound probe was utilized to scan and analyze skin collagen density. Units: Intensity score

SECONDARY OUTCOMES:
The change of skin texture | Change from Baseline skin texture at 4 weeks
  VISIA Complexion Analysis System was utilized to measure skin texture. Units: arbitrary units
The change of skin pores | Change from Baseline skin pores at 4 weeks
  VISIA Complexion Analysis System was utilized to measure skin pores. Units: arbitrary units

CONTACTS AND LOCATIONS:
Overall Officials: Chia-Hua Liang, Principal Investigator — Chia Nan University of Pharmacy ＆ Science
Locations (1):
- Chia Nan University of Pharmacy ＆ Science, Tainan, Taiwan